CLINICAL TRIAL: NCT00356122
Title: A Phase II Multicenter Study of Docetaxel and Oxaliplatin in Combination With Bevacizumab as First-Line Treatment in Chemotherapy-Naïve Subjects With Unresectable Locally Advanced and/or Recurrent (Stage IIIB) or Metastatic (Stage IV) Non-Squamous Cell Histology Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Docetaxel & Oxaliplatin in Combination With Bevacizumab as First-Line Treatment in Subjects With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCOX_L_00716
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung; non-small cell; chemotherapy; tumor; advanced; recurrent; metastatic; Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Docetaxel; Oxaliplatin; Bevacizumab

ARMS (1):
- Docetaxel/Oxaliplatin/Bevacizumab (Experimental): Participants with advanced, recurrent, or metastatic Non Small Cell Lung Cancer (NSCLC), treated with the combination of docetaxel, followed by oxaliplatin, and then bevacizumab for Cycles 1-6 (every 3 weeks), and followed with maintenance therapy with bevacizumab every 3 weeks for a total of 52 weeks.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — 70 mg/m^2 administered intravenously (IV) on Day 1 for Cycles 1-6 (the treatment cycle is 3 weeks)
Drug: Oxaliplatin — 100 mg/m^2 administered IV on Day 1 for Cycles 1-6
Drug: Bevacizumab — 15 mg/kg administered IV on Day 1 for Cycles 1-6, and every 3 weeks during maintenance therapy for a total treatment of one year, until disease progression or death due to any cause, whichever occurs first.

SUMMARY:
The purpose of this study was to see how well three investigational drugs worked together in preventing progression of the disease. This study provided a new combination of chemotherapy drugs - docetaxel and oxaliplatin - as first line therapy in the treatment of lung cancer. The therapy included bevacizumab that may prevent or slow down the blood supply to the tumor and may also prevent tumor growth. The three investigational drugs are United States Food and Drug Administration (FDA) approved.

DETAILED DESCRIPTION:
The planned treatment duration for each participant is six 21-day treatment cycles of combination therapy; non-progressing participants will continue on bevacizumab monotherapy until progression. After discontinuation or after completion of all study treatments, all participants will be contacted every 3 months for a maximum of 2 years from first treatment to document overall survival and record new anticancer treatment (chemotherapy or biologic).

ELIGIBILITY:
Inclusion Criteria

Participants who met all of the following criteria during screening were considered for enrollment into the study:

1. Had the informed consent in writing for all prior to registration into the study
2. Had histologic or cytologic confirmation of locally advanced or metastatic (stage IIIb/IV) NSCLC (non-squamous histology). Participants with mixed tumor types could have been enrolled, unless small cell elements were discovered
3. Had measurable disease, defined as at least 1 lesion that could be accurately measured in at least 1 dimension (longest diameter) as ≥ 2.0 cm with conventional computerized tomography (CT) or magnetic resonance imaging (MRI) scans, or as ≥ 1.0 cm with spiral CT scan
4. Had no prior systemic chemotherapy
5. Was male or female ≥ 18 years old
6. Had an estimated life expectance of ≥ 12 weeks
7. Had an ECOG performance status (PS) of 0, 1, or 2
8. Was a nonpregnant, nonlactating female Was a male or female of childbearing potential who was willing to use an effective form of contraception while on therapy and for 90 days thereafter.
9. Had adequate renal function as determined by the following within 2 weeks prior to study registration.

   * A calculated creatinine clearance greater than 45 mL/min using the Cockcroft-Gault formula
   * A urine dipstick or urinalysis for protein <2+ (Participants discovered to have ≥ 2+ proteinuria on dipstick or urinalysis at baseline had to undergo a 24 hour urine collection and had to have ≤ 1 gm of protein over 24 hours to be eligible).
10. Had a hematologic evaluation within 2 weeks prior to study registration (and met the minimum values):

    * Had absolute neutrophil count (ANC) ≥ 1,500 cells/microL
    * Had platelet count ≥ 100,000 cells/microL
    * Had hemoglobin ≥ 9.9 gm/deciL (erythropoietin [e.g., Epogen®] could have been used to maintain or exceed this level)
    * Had a partial thromboplastin time (PTT) ≤ upper limit of normal (ULN)
11. Had a hepatic function evaluation within 2 weeks prior to study registration met the eligibility criteria for bilirubin, Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase.

Exclusion criteria

Participants with any of the following were not included in the study:

1. Had received prior systemic chemotherapy or vascular endothelial growth factor (VEGF) or epidermal growth factor receptor (EGFR) inhibitor therapy at any time; or had received recent or current radiation therapy
2. Had intrathoracic lung carcinoma of squamous cell histology. (Participants with extrathoracic-only squamous cell NSCLC were eligible. Participants with only peripheral lung lesions (of any NSCLC histology) were also eligible
3. Had cardiovascular diseases and related treatment, including the following:

   * New York Heart Association Class ≥ 2 congestive heart failure; participants with a history of serious cardiac disease not adequately controlled; or a history of myocardial infarction or unstable angina pectoris within 6 months prior to study registration
   * History of stroke or transient ischemic attack within 6 months of study registration
   * History of hypertensive crisis or hypertensive encephalopathy
   * History of thrombotic or hemorrhagic disease
   * Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
   * Clinically meaningful peripheral vascular disease, or arrhythmia
   * Inadequately controlled blood pressure (defined as systolic blood pressure >150 mm Hg and/or diastolic blood pressure >100 mm Hg)
   * Significant vascular disease (e.g., aortic aneurysm, aortic dissection) within 6 months prior to study registration
   * Therapeutic anticoagulation (Participants receiving prophylactic anticoagulation for venous access devices were allowed providing they met certain criteria)
   * Chronic daily treatment with aspirin (≥ 325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function; treatment with dipyridamole, ticlopidine, clopidogrel, or cilostazol was not allowed.
4. Had a surgical procedure in anamnesis (medical history):

   * Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to study registration, or anticipation of need for major surgical procedure during the course of the study
   * In the case of high-risk procedures, such as liver resection, thoracotomy, or neurosurgery, within 8 weeks prior to study registration
   * Minor surgical procedures (e.g., fine needle aspirations, core biopsies) within 7 days prior to registration
5. Had a serious nonhealing wound, active ulcer, or untreated bone fracture
6. Had a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study registration
7. Had a history of gross hemoptysis (defined as bright red blood of ≥ 0.5 teaspoon) within 4 weeks prior to study registration
8. Had a history of hypersensitivity reaction to drugs formulated with polysorbate 80 or platinum containing compounds
9. Had peripheral neuropathy ≥ Grade 2 (based on CTCAE v3.0)
10. Had known central nervous system (CNS) disease, except for treated brain metastasis. However, participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to study registration were excluded.
11. Had a history of a malignancy other than NSCLC; exceptions to this included:

    * Curatively treated basal cell carcinoma, cervical intraepithelial neoplasia, or localized prostate cancer with a current prostate-specific antigen (PSA) of less than 1.0 ng/dL on 2 successive evaluations at least 3 months apart, and the most recent evaluation being within 4 weeks of study registration
    * History of another malignancy that was curatively treated and no evidence of disease for a minimum of 5 years
12. Had symptoms of a clinically meaningful illness in the 90 days before study registration, or had history of other disease, (such as human immunodeficiency virus [HIV] positive, chronic infection [e.g., pulmonary tuberculosis], or hepatitis A, B, or C [active or previously treated]), had an active infection with fever, had metabolic dysfunction, had physical examination finding, or had clinical a laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug, that might affect the interpretation of the results of the study, or render the participant at high risk from treatment complications; (testing for these conditions was at investigator discretion)
13. Had a mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study

The above information is not intended to contain all considerations relevant to a patients potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Erickson, MSN, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in 18 sites in the United States, of which 14 sites enrolled a total of 85 participants.
Pre-assignment Details: Of the 85 participants screened for this study, 32 were screen-failures. 53 participants were registered to receive treatment in this study, however, one participant did not receive any study medication.
  All 53 participants entered the follow-up period, even if they discontinued treatment.
Groups:
- Docetaxel/Oxaliplatin/Bevacizumab: Participants with advanced, recurrent, or metastatic Non Small Cell Lung Cancer (NSCLC), treated with the combination of
  * 70 mg/m^2 docetaxel intravenously on Day 1 for Cycles 1-6,
  * 100 mg/m^2 oxaliplatin intravenously on Day 1 for Cycles 1-6,
  * 15 mg/kg bevacizumab intravenously on Day 1 for Cycles 1-6 and every 3 weeks during maintenance therapy.
Period: TREATMENT
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Started | 53
Completed | 8
Not Completed | 45
Not completed — Lack of Efficacy | 26
Not completed — Adverse Event | 10
Not completed — Subject's request | 4
Not completed — Other | 4
Not completed — Did not receive study medication | 1
Period: FOLLOW-UP
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Started | 53
Completed | 12
Not Completed | 41
Not completed — Death | 37
Not completed — Lost to Follow-up | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 61.10 (11.07)
Age, Customized [Number; unit: participants]
  <65 years | 28
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 38
Weight [Mean (Standard Deviation); unit: kilograms] | 76.530 (17.793)
Height [Mean (Standard Deviation); unit: Centimeters] | 169.80 (9.57)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: Square meters] — BSA was calculated using the Mosteller formula if it was missing
  Square meters | 1.875 (0.252)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from the date of registration to the earliest date of documented evidence of progressive disease, or the date of death due to any cause, whichever occurred first.
  Progressive disease occurred when the participant had at least a 20% increase in the sum of the longest diameter (LD) of target lesions, compared to the smallest sum LD recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: Baseline to PFS (up to 24 months after the first treatment)
Population: All participants registered to receive study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 53
Months | 5.6 [3.7 to 7.6]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate is the percentage of participants with an objective response. Improvements in tumor measurements from baseline values were assigned a status of Complete Response (CR) or Partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST). Overall objective response was the sum of CR and PR.
  CR referred to the disappearance of all target lesions, and PR was at least 30% decrease in the sum of the longest diameter (LD) of target lesions, compared to the baseline sum LD. Responses were confirmed by repeat assessments within 4 to 6 weeks.
Time Frame: Baseline to CR or PR (up to 24 months after the first treatment)
Population: All participants registered to receive study treatment
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 53
Percentage of participants | 30.2 [18.3 to 44.3]

3. Secondary Outcome: Time-to-treatment Failure (TTF)
Description: Treatment failure was defined as an event which lead to the participant's withdrawal from the study treatment due to lack of efficacy, disease progression, adverse events, or due to a participant's request as recorded in the Case Report Form (CRF), death, or use of other anticancer therapy.
  TTF was assessed using Kaplan-Meier method, and the median TTF with 95% CIs was computed using the Brookmeyer and Crowley method.
Time Frame: Baseline to treatment failure (up to 24 months after the first treatment)
Population: All participants registered to receive study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 53
Months | 4.7 [2.9 to 5.6]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from the date of registration to the date of death due to any cause, or to the date of last contact (for censored observations). OS was assessed by the Kaplan-Meier method and the estimates of median survival time with 95% CI are reported.
Time Frame: Baseline to OS (up to 24 months after the first treatment)
Population: All participants registered to receive study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 53
Months | 14.0 [9.9 to 16.9]

5. Secondary Outcome: Number of Participants With Treatment-related Toxicities
Description: Treatment-related toxicities were serious and non-serious adverse events (AE) considered related to study treatment by the investigator.
  AEs were any unfavorable and unintended signs, symptoms, syndromes, or illnesses that developed or worsened during the observation period, and included abnormal results from diagnostic procedures. Serious AEs resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability or incapacity, appeared as a congenital anomaly or were considered medically important by the investigator.
Time Frame: From baseline up to 30 days after treatment discontinuation
Population: All participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Number analyzed (Participants) | 52
Participants
  At least one AE related to docetaxel | 51
  At least one AE related to oxaliplatin | 50
  At least one AE related to bevacizumab | 43

ADVERSE EVENTS:
Description: In the table below for 'other adverse events', the number of participants affected are participants who exhibited one or more of any adverse event.
Arm/Group | Docetaxel/Oxaliplatin/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 17/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Oxaliplatin/Bevacizumab (N=52)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 2
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 1
PNEUMONIA (Infections and infestations) | 4
SEPSIS (Infections and infestations) | 2
APPENDICITIS (Infections and infestations) | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 1
WRONG DRUG ADMINISTERED (Injury, poisoning and procedural complications) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
OESOPHAGOBRONCHIAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Oxaliplatin/Bevacizumab (N=52)
NEUTROPENIA (Blood and lymphatic system disorders) | 10
LEUKOPENIA (Blood and lymphatic system disorders) | 7
ANAEMIA (Blood and lymphatic system disorders) | 5
DIARRHOEA (Gastrointestinal disorders) | 33
NAUSEA (Gastrointestinal disorders) | 32
VOMITING (Gastrointestinal disorders) | 21
CONSTIPATION (Gastrointestinal disorders) | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 10
STOMATITIS (Gastrointestinal disorders) | 10
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
HAEMORRHOIDS (Gastrointestinal disorders) | 4
DYSPEPSIA (Gastrointestinal disorders) | 3
DYSPHAGIA (Gastrointestinal disorders) | 3
FATIGUE (General disorders) | 37
PYREXIA (General disorders) | 12
MUCOSAL INFLAMMATION (General disorders) | 6
CHILLS (General disorders) | 4
NON-CARDIAC CHEST PAIN (General disorders) | 4
ASTHENIA (General disorders) | 3
HYPERSENSITIVITY (Immune system disorders) | 5
FUNGAL INFECTION (Infections and infestations) | 4
URINARY TRACT INFECTION (Infections and infestations) | 3
WEIGHT DECREASED (Investigations) | 11
HAEMOGLOBIN DECREASED (Investigations) | 5
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5
NEUTROPHIL COUNT DECREASED (Investigations) | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 3
PLATELET COUNT DECREASED (Investigations) | 3
ANOREXIA (Metabolism and nutrition disorders) | 15
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 9
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 8
DEHYDRATION (Metabolism and nutrition disorders) | 7
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
DYSGEUSIA (Nervous system disorders) | 10
NEUROPATHY PERIPHERAL (Nervous system disorders) | 10
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 9
HEADACHE (Nervous system disorders) | 7
INSOMNIA (Psychiatric disorders) | 14
DEPRESSION (Psychiatric disorders) | 6
ANXIETY (Psychiatric disorders) | 5
PROTEINURIA (Renal and urinary disorders) | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 12
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 5
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 5
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 24
RASH (Skin and subcutaneous tissue disorders) | 5
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 4
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 3
HYPERTENSION (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 60 days in advance of any submission for publication. The Sponsor may request for the publication to be delayed for a limited time, not to exceed 90 days to preserve its proprietary rights.